CLINICAL TRIAL: NCT00806351
Title: Efficacy And Safety Of Eraxis/Ecalta (Anidulafungin) Compared To Cancidas (Caspofungin) In Neutropenic Patients With Invasive Candida Infection
Brief Title: An Evaluation Of The Effectiveness And Safety Of Anidulafungin Compared To Caspofungin For The Treatment Of Serious Fungal Infection Due To Candida In Patients With A Dysfunctional Immune System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was prematurely terminated on May 18, 2012 due to slow enrollment. The study was not terminate due to any safety issues or concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8851021
Record Dates: First submitted 2008-11-26; First posted 2008-12-10 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-11

CONDITIONS: Fungemia; Neutropenia; Candidiasis
Keywords: Candidiasis; Invasive Candidiasis; Candida; Candidemia; Fungal Infection; Neutropenia
MeSH Terms: conditions — Fungemia; Neutropenia; Candidiasis; Candidiasis, Invasive; Torulopsis; Candidemia; Mycoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anidulafungin Arm (Experimental): Subjects were randomized 2:1 (anidulafungin:caspofunin).
  Interventions: Drug: Active Anidulafungin
- Caspofungin Arm (Experimental): Subjects were randomized 2:1 (anidulafungin:caspofunin).
  Interventions: Drug: Active Caspofungin

INTERVENTIONS:
Drug: Active Anidulafungin — Subjects in this arm will receive active anidulafungin and placebo caspofungin
  Arms: Anidulafungin Arm
Drug: Active Caspofungin — Subjects in this arm will receive active caspofungin and placebo anidulafungin
  Arms: Caspofungin Arm

SUMMARY:
The purpose of this study is to gather information on the use of anidulafungin for the treatment of Candida infection in patients with an abnormal immune system. It is expected that anidulafungin will be at least as safe and as effective as the comparator drug, caspofungin.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional immune system (reduced neutrophils).
* Confirmed Candida infection, defined as growth of Candida from a normally sterile site accompanied by signs and symptoms of infection.
* Male of female ≥16 years of age.
* Expected hospitalization for at least ten (10) days.

Exclusion Criteria:

* Pregnancy or breast feeding or planning to become pregnant during the study.
* Recent treatment with one of the study drugs over the last 30 days.
* Allergy to either study drug or to this class of drugs.
* Significant liver dysfunction.
* Suspected Candida osteomyelitis, endocarditis, meningitis or any other infections of the central nervous system.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Pfizer Investigational Site, Sarajevo, Bosnia and Herzegovina
- France (2):
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Strasbourg
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Roma
- Poland (3):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Košice, Slovakia

REFERENCES:
- [Derived] De Rosa FG, Busca A, Capparella MR, Yan JL, Aram JA. Invasive Candidiasis in Patients with Solid Tumors Treated with Anidulafungin: A Post Hoc Analysis of Efficacy and Safety of Six Pooled Studies. Clin Drug Investig. 2021 Jun;41(6):539-548. doi: 10.1007/s40261-021-01024-7. Epub 2021 Apr 23. PMID 33891293
- [Derived] Kontoyiannis DP, Bassetti M, Nucci M, Capparella MR, Yan JL, Aram J, Hogan PA. Anidulafungin for the treatment of candidaemia caused by Candida parapsilosis: Analysis of pooled data from six prospective clinical studies. Mycoses. 2017 Oct;60(10):663-667. doi: 10.1111/myc.12641. Epub 2017 Jun 9. PMID 28597967
- [Derived] Kullberg BJ, Vasquez J, Mootsikapun P, Nucci M, Paiva JA, Garbino J, Yan JL, Aram J, Capparella MR, Conte U, Schlamm H, Swanson R, Herbrecht R. Efficacy of anidulafungin in 539 patients with invasive candidiasis: a patient-level pooled analysis of six clinical trials. J Antimicrob Chemother. 2017 Aug 1;72(8):2368-2377. doi: 10.1093/jac/dkx116. PMID 28459966
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851021&StudyName=An%20Evaluation%20Of%20The%20Effectiveness%20And%20Safety%20Of%20Anidulafungin%20Compared%20To%20Caspofungin%20For%20The%20Treatment%20Of%20Serious%20Fungal%20Infection%20Due

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: Participants received anidulafungin (100 milligrams [mg]) followed by matched placebo-caspofungin once daily (QD) or participants received matched placebo-caspofungin followed by active anidulafungin (100 mg) QD. Anidulafungin loading dose on Day 1 was 200 mg. Study treatments given either entirely as intravenous (IV) therapy or if protocol-specified criteria met, as sequential IV (at least 10 days) then oral antifungal therapy (14 days). Dosage of antifungal therapy (fluconazole or voriconazole tablets) determined by the Investigator. A maximum of 42 days of IV study treatment and a maximum of 14 days of oral study treatment allowed. Thus, participants may have received up to a maximum of 56 days of study therapy.
- Caspofungin: Participants received caspofungin (35, 50, or 70 mg depending on participant's weight, baseline liver function, or receipt of an interacting drug) followed by matched placebo-anidulafungin QD or participants received matched placebo-anidulafungin followed by active caspofungin (35, 50, or 70 mg) QD. Caspofungin loading dose on Day 1 was 70 mg. Study treatments given either entirely as IV therapy or if protocol-specified criteria met, as sequential IV (at least 10 days) then oral antifungal therapy (14 days). Dosage of antifungal therapy (fluconazole or voriconazole tablets) determined by the Investigator. A maximum of 42 days of IV study treatment and a maximum of 14 days of oral study treatment allowed. Thus, participants may have received up to a maximum of 56 days of study therapy.
Period: Overall Study
Arm/Group | Anidulafungin | Caspofungin
Started | 15 | 6
Completed | 10 | 2
Not Completed | 5 | 4
Not completed — Death | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anidulafungin | Caspofungin | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Customized [Number; unit: participants]
  18 to 44 years | 2 | 2 | 4
  45 to 64 years | 9 | 2 | 11
  greater than or equal to (≥) 65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Global Response at End of Intravenous Treatment (EOIVT)
Description: Participant counts of global response of success, failure, or indeterminate. Success: clinical response of cure (no signs, symptoms [s/s] of Candida) or improvement (significant, incomplete resolution of s/s) and microbiological response of eradication (follow-up [f/u] culture negative) or presumed eradication (f/u culture not available and clinical success). Failure: clinical response of failure (greater than or equal to [≥3] doses study medication and no significant improvement of s/s or death due to Candida) and/or unsuccessful microbiological response of persistent(positive culture any Candida species [sp]), new infection or relapse at f/u. Indeterminate: clinical and/or microbiological response of indeterminate (evaluation could not be made due to withdrawal from study prior to assessment of cure or failure) and there was neither clinical response of failure nor unsuccessful microbiological response (persistence or new infection or relapse).
Time Frame: Day 10 up to Day 42
Population: Modified Intent to Treat (MITT) Population: participants who received at least 1 dose of study medication and had positive culture for Candida sp isolated from cultures obtained from a normally sterile site within 96 hours prior to treatment initiation. A global response of failure at EOIVT was carried forward programmatically to subsequent visits.
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 11 | 3
participants
  Success | 8 | 3
  Failure | 3 | 0
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; The 95 percent confidence interval (95% CI) was calculated using the method of exact unconditional confidence limits for the difference. Global response (rates of success) by using a 2-sided 95% CI for the true difference in efficacy (Anidulafungin minus Caspofungin) was calculated. Statistical testing was done at 2.5% alpha; Test type: Superiority or Other; Risk Difference = -27.3, 95% CI 2-sided [-80.9 to 40.3]

2. Secondary Outcome: Global Response at End of Treatment (EOT)
Description: Participant counts of global response of success, failure, or indeterminate. Success: clinical response of cure (no s/s of Candida) or improvement (significant, incomplete resolution of s/s) and microbiological response of eradication (f/u culture negative) or presumed eradication (f/u culture not available and clinical success). Failure: clinical response of failure (≥3 doses study medication and no significant improvement of s/s or death due to Candida) and/or unsuccessful microbiological response of persistent (positive culture any Candida sp), new infection or relapse at f/u. Indeterminate: clinical and/or microbiological response of indeterminate (evaluation could not be made due to withdrawal from study prior to assessment of cure or failure) and there was neither clinical response of failure nor unsuccessful microbiological response (persistence or new infection or relapse).
Time Frame: Day 14 up to Day 56
Population: MITT Population; A global response of failure at EOT was carried forward programmatically to all subsequent visits.
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 11 | 3
participants
  Success | 8 | 3
  Failure | 3 | 0
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; The 95% CI was calculated using the method of exact unconditional confidence limits for the difference. Global response (rates of success) by using a 2-sided 95% CI for the true difference in efficacy (Anidulafungin minus Caspofungin) was calculated. Statistical testing was done at 2.5% alpha; Test type: Superiority or Other; Risk Difference = -27.3, 95% CI 2-sided [-80.9 to 40.3]

3. Secondary Outcome: Global Response at 2-Week Follow-Up Visit
Description: as for outcome 2
Time Frame: 2 weeks post treatment
Population: MITT Population; subset of participants who, according to the investigator, completed therapy and participants with global response of failure at EOIVT or EOT. A global response of failure at the 2-week and 6-week visits carried forward programmatically to all subsequent visits. Number of participants analyzed (N): participants with evaluable data.
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 9 | 1
participants
  Success | 6 | 1
  Failure | 3 | 0
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Risk Difference = -40.0, 95% CI 2-sided [-97.5 to 63.9]

4. Secondary Outcome: Global Response at 6-Week Follow-Up Visit
Description: as for outcome 2
Time Frame: 6 weeks post treatment
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 9 | 1
participants
  Success | 5 | 1
  Failure | 4 | 0
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Risk Difference = -50.0, 95% CI 2-sided [-97.5 to 55.0]

5. Secondary Outcome: Response Based on Clinical Cure and Microbiological Success at EOIVT
Description: Participant counts of clinical cure (no s/s of Candida) and microbiological success (eradication [f/u culture negative] or presumed eradication [f/u culture not available and a clinical response of cure]).
Time Frame: Day 10 up to Day 42
Population: MITT Population; subset of participants with clinical cure or improvement and microbiological eradication or presumed eradication. A global response of failure at EOIVT was carried forward programmatically to all subsequent visits.
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 8 | 3
participants | 7 | 2

6. Secondary Outcome: Response Based on Clinical Cure and Microbiological Success at EOT
Description: as for outcome 5
Time Frame: Day 14 up to Day 56
Population: MITT Population; subset of participants with clinical cure or improvement and microbiological eradication or presumed eradication. A global response of failure at EOT was carried forward programmatically to all subsequent visits.
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 8 | 3
participants | 6 | 3

7. Secondary Outcome: Response Based on Clinical Cure and Microbiological Success at 2-Week Follow-Up Visit
Description: as for outcome 5
Time Frame: 2 weeks post treatment
Population: MITT Population; subset of participants with clinical cure or improvement and microbiological eradication or presumed eradication; Number of participants analyzed (N): participants with evaluable data a specified time point
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 6 | 1
participants | 4 | 1

8. Secondary Outcome: Response Based on Clinical Cure and Microbiological Success at 6-Week Follow-Up Visit
Description: as for outcome 5
Time Frame: 6 weeks post treatment
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 6 | 1
participants | 6 | 1

9. Secondary Outcome: Clinical Response at Day 10
Description: Participant counts of clinical response categorized as success, failure, or indeterminate. Success: no s/s of Candida (cure) or significant but incomplete resolution of s/s of Candida; no additional systemic or oral antifungal treatment required (improvement). Failure: worsening of s/s of the Candida infection. Indeterminate: evaluation could not be made due to withdrawal from study prior to assessment of cure or failure. Participants who received fewer than 3 doses of study medication were assigned a clinical efficacy response of indeterminate.
Time Frame: Day 10
Population: MITT Population; Number of participants analyzed (N): participants with evaluable data
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 9 | 3
participants
  Success | 7 | 3
  Failure | 0 | 0
  Indeterminate | 2 | 0
Statistical Analysis 1: Comparison: Anidulafungin vs Caspofungin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Risk Difference = -36.4, 95% CI 2-sided [-90.6 to 31.9]

10. Secondary Outcome: Number of Participants With Recurrence
Description: Participant counts of microbiologic response of recurrence defined as any baseline Candida sp isolated following eradication, or culture data were not available for participants with a clinical response of failure after a previous response of success. Clinical failure defined as ≥3 doses study medication and no significant improvement of s/s or death due to Candida. Clinical success is resolution of s/s and no additional antifungal treatment needed.
Time Frame: 2 and 6 weeks post treatment
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 11 | 3
participants
  2 Weeks post treatment | 0 | 0
  6 Weeks post treatment | 0 | 0

11. Secondary Outcome: Number of Participants With New Infections
Description: Participant counts of microbiologic response of new infection defined as clinical failure with emergence of new Candida sp not identified at baseline at the original site of infection or at a distant site of infection. Clinical failure defined as ≥3 doses study medication and no significant improvement of s/s or death due to Candida.
Time Frame: 2 and 6 weeks post treatment
Population: MITT Population
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 11 | 3
participants
  2 weeks post treatment | 0 | 0
  6 weeks post treatment | 0 | 0

12. Secondary Outcome: Time to First Negative Blood Culture for Candida Species
Description: A participant had a negative blood culture, if having determined the day of the first negative blood culture, the subsequent blood culture was also negative, or if positive, the interval between the cultures was at least 2 days. For participants whose blood culture went from positive to negative, the time to negative blood culture defined as: date of first negative blood culture minus first treatment date plus 1.
Time Frame: Baseline up to Day 56
Population: MITT Population; subset of participants who had a positive blood culture for Candida sp. on Day 1 of treatment. No participant in the Caspofungin treatment arm had a positive blood culture for Candida sp. on Day 1 of treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 5
days | 2.0 [2 to 5]

13. Secondary Outcome: Time to Death
Description: Time to death defined as: date of death minus first treatment date plus 1.
Time Frame: Day 1 up to Day 98
Population: Safety Population;subset of participants who died
Measure: Median (Full Range); unit: days
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 5 | 4
days | 34.0 [5 to 36] | 15.5 [3 to 41]

14. Secondary Outcome: All-Cause Mortality
Description: All-cause mortality during study therapy and at follow-up visits reported as unique deaths at EOIVT, end of oral treatment (EOT-oral), 2 Week Follow-Up and 6 Week Follow-Up
Time Frame: Baseline up to 6 weeks post treatment
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Caspofungin
Number analyzed (Participants) | 15 | 6
participants
  at EOIVT | 1 | 1
  at EOT - oral | 1 | 0
  at 2 Week Follow-Up Visit | 1 | 3
  at 6 Week Follow-Up Visit | 2 | 0

ADVERSE EVENTS:
Description: All-causality events reported. The same event may appear as both an adverse event (AE) and serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin | Caspofungin
Serious Adverse Events (participants affected / at risk) | 5/15 | 4/6
Other Adverse Events (participants affected / at risk) | 14/15 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=15) | Caspofungin (N=6)
Drug ineffective (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=15) | Caspofungin (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Colour blindness acquired (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Phosphenes (Eye disorders) | 0 | 1
Retinal exudates (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Visual brightness (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gingival disorder (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Aspergillosis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 2 | 0
Furuncle (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Bacterial test positive (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Fungal test positive (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Weight increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Costovertebral angle tenderness (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hyperaemia (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Palatal disorder (Gastrointestinal disorders) | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study prematurely terminated due to slow enrollment, not due to safety issues. Meaningful interpretation and comparison of treatment outcomes with caspofungin was difficult due to low number of participants (n=3) with confirmed Candida infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.